CLINICAL TRIAL: NCT02186964
Title: Randomised Prospective Comparison of Tension-free Primary Closure, Karydakis and Limberg Flap Methods in Treatment of Pilonidal Sinus Disease
Brief Title: Comparison of Tension Free Primary Closure, Karydaks and Limberg Flap Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, barış sevinç, MD, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS42
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Pilonidal Disease; Recurrence; Complication
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- tension free primary closure (Experimental): patients treated by tension free primary closure
  Interventions: Procedure: tension free primary closure
- karydakis (Experimental): patients treated by Karydakis method
  Interventions: Procedure: karydakis
- Limberg flap (Experimental): patients treated by Limberg flap procedure
  Interventions: Procedure: Limberg flap

INTERVENTIONS:
Procedure: tension free primary closure — tension free primary closure of the defects created by excision of the pilonidal sinus
  Arms: tension free primary closure
Procedure: karydakis — the defect after excision of the pilonidal sinus is closed by Karydakis procedure
  Arms: karydakis
Procedure: Limberg flap — defect after excision of the pilonidal sinus is closed by Limberg flap procedure
  Arms: Limberg flap

SUMMARY:
Pilonidal sinus is a chronic inflammatory disorder of intergluteal sulcus. The disease seen in between 15-35 years of age and 3-4 times more in males. The incidence of the disease is found as 8.8% in Turkish soldiers. The disorder mainly affects the quality of life.

There are numerous methods in surgical treatment of Pilonidal sinus. The main difference in between those methods is the closing of the defect that occurs after the excision of the sinus tract. The defect can be closed by primary sutures or it can be left for secondary healing. Nowadays, the recurrence rate of flap procedures are lower therefore, flap procedures are commonly used. However, it has been reported that there is no difference between flap procedures and tension free primary closure. This result triggered the controversy that; if the healing side is tension free, midline suturing may have no importance. The aim of this study is to compare the results of 3 different surgical procedures used in treatment of pilonidal disease.

ELIGIBILITY:
Inclusion Criteria:

* having pilonidal sinus disease
* desire for surgical treatment
* accept to be involved in the study

Exclusion Criteria:

* patients under age of 18
* recurrent cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
recurrence | 2 years
  recurrence rates two years after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Karahan, Professor, Study Director — Konya Meram State Hospital
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Sevinc B, Karahan O, Okus A, Ay S, Aksoy N, Simsek G. Randomized prospective comparison of midline and off-midline closure techniques in pilonidal sinus surgery. Surgery. 2016 Mar;159(3):749-54. doi: 10.1016/j.surg.2015.09.024. Epub 2015 Oct 31. PMID 26531235